CLINICAL TRIAL: NCT02676115
Title: The Use of Wound Taping Protocol to Improve Cosmetic Scar After Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: Medipore Tape Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-00048
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Scarring
Keywords: Cosmetic Wound Healing; anterior cruciate ligament (ACL)
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Standard Post Operative Skin Care
  Interventions: Other: Standard Post Operative Skin Care
- Treatment Group (Experimental): Medipore Tape will be applied to ACL reconstruction Incision
  Interventions: Other: Medipore Tape

INTERVENTIONS:
Other: Standard Post Operative Skin Care — Control group subjects will receive the standard post-operative skin care which are steri-strips covered with gauze, and this will be removed at the first visit. No additional skin dressings will be used in the control group.
  Arms: Control Group
Other: Medipore Tape — * One layer of Medipore tape will be placed across the incision.
  * Patients will be instructed on how to change the tape, and will be encouraged to change the tape as often as once per week for hygiene.
  When patients return to the office for their regularly scheduled visit, the Medipore tape will be changed and a picture of the scar will be taken.
  Arms: Treatment Group

SUMMARY:
This is a prospective, single-blinded, two-arm, randomized, parallel, pragmatic, effectiveness trial that will enroll patients undergoing arthroscopic anterior cruciate ligament reconstruction in order to evaluate the efficacy of using Medipore tape to improve cosmetic wound healing and scaring.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing arthroscopic ACL reconstruction with bone-patella-tendon-bone autograft at the Ambulatory Surgical Center and Hospital for Joint Diseases will be eligible for enrollment.
* Patient is indicated for ACL reconstructive surgery with bone-patella-tendon-bone autograft

Exclusion Criteria:

* Subjects/Parents who are mentally impaired and are unable to give consent
* Patients with prior vertical anterior knee incisions
* Patients with known skin reactions to adhesive
* Patients with high risk for abnormal scar formation and keloids

Ages: 15 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in patients' own appraisal of their scar assessed quantitatively by change in Manchester Scar Scale (MSS) Score | 6 Months
Quantitative Assessment of Scar using Patient and Observer Scar Assessment Scale (POSAS) | 6 Months
Dermatology Life Quality Index (DLQI) | 6 Months
  Quantitative assessment of health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States